CLINICAL TRIAL: NCT02953509
Title: A Phase 1b/2 Trial of Hu5F9-G4 in Combination With Rituximab or Rituximab + Chemotherapy in Patients With Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Brief Title: Trial of Magrolimab (Hu5F9-G4) in Combination With Rituximab or Rituximab + Chemotherapy in Participants With Relapsed/Refractory B-cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to the magrolimab program discontinuation.
Sponsor: Gilead Sciences (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5F9003; 2016-003408-29 (EudraCT Number)
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — magrolimab; Rituximab; Gemcitabine; Oxaliplatin; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab (Experimental): Participants with B-cell non-hodgkin's lymphoma (NHL) will receive 1 mg/kg magrolimab intravenous (IV) infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 10 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Each cycle length of 28 days.
  Interventions: Drug: Magrolimab; Drug: Rituximab
- Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab (Experimental): Participants with B-cell NHL will receive 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 20 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Each cycle length of 28 days.
  Interventions: Drug: Magrolimab; Drug: Rituximab
- Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab (Experimental): Participants with B-cell NHL will receive 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11,15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Each cycle length of 28 days.
  Interventions: Drug: Magrolimab; Drug: Rituximab
- Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab (Experimental): Participants with B-cell NHL will receive 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Each cycle length of 28 days.
  Interventions: Drug: Magrolimab; Drug: Rituximab
- Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin (Experimental): Autologous stem cell transplant ineligible diffuse large B-cell lymphoma (DLBCL) participants will receive 1 mg/kg magrolimab IV infusion priming dose(over 3 hours)on Day 1 of Cycle 1,followed by maintenance dose of 30 mg/kg on Days 8, 11, 15, 22, and 29 of Cycle 1;Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles.Cycle length will be 28 days.Rituximab 375 mg/m^2 IV infusion will be given on Days 8, 15, 22, and 29 of Cycle 1,followed by 1 dose on Day 1 of Cycles 2 to 6.Thereafter from Cycle 8 and beyond,rituximab will be administered on Day 1 of every other cycle(on even cycles).Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion will be given as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4.Granulocyte colony stimulating factor (G-CSF) prophylaxis will be given with gemcitabine and oxaliplatin treatment(Cycles 1-4).Allopurinol 300 mg orally daily will be administered for the first cycle only.
  Interventions: Drug: Magrolimab; Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Allopurinol
- Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin (Experimental): Autologous stem cell transplant ineligible DLBCL participants will receive 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 45 mg/kg on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length of 28 days. Rituximab 375 mg/m^2 IV infusion will be administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion will be administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis will be administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily will be administered for the first cycle only.
  Interventions: Drug: Magrolimab; Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Allopurinol
- Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab (Experimental): Participants with B-cell indolent NHL (iNHL) (including follicular lymphoma [FL] and marginal zone lymphoma [MZL]) and DLBCL will receive 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Each cycle length of 28 days.
  Interventions: Drug: Magrolimab; Drug: Rituximab
- Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab (Experimental): Participants with B-cell iNHL (including FL and MZL) and DLBCL will receive 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, and 22 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Each cycle length of 28 days.
  Interventions: Drug: Magrolimab; Drug: Rituximab
- Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab (Experimental): Participants with B-cell iNHL (including FL and MZL) and DLBCL will receive 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, and 22 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Each cycle length of 28 days.
  Interventions: Drug: Magrolimab; Drug: Rituximab
- Phase 2 Cohort 4: Magrolimab 30 mg/kg + Rituximab (Experimental): Participants with DLBCL will receive 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab will be administered on Day 1 of every other cycle (on even cycles). Each Cycle length of 28 days.
  Interventions: Drug: Magrolimab; Drug: Rituximab

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: Hu5F9-G4
Drug: Rituximab — Administered intravenously on Days 8, 15, and 22 during Cycle 1, followed by 1 dose on Day 1 for Cycles 2 through 6, and Day 1 for every other cycle until Cycle 13
  Other Names: RITUXAN®; MabThera
Drug: Gemcitabine — Administered intravenously on Days 11, 23 for Cycle 1 and Days 2 and 15 for Cycles 2 to 4
  Other Names: Gemzar®
  Arms: Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin; Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Drug: Oxaliplatin — Administered intravenously on Days 11, 23 for Cycle 1 and Days 2 and 15 for Cycles 2 to 4
  Other Names: Eloxatin®
  Arms: Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin; Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Drug: Allopurinol — Administered orally during Cycle 1
  Arms: Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin; Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin

SUMMARY:
The primary objectives of this study are:

* To investigate the safety and tolerability, and to define the recommended Phase 2 dose and schedule (RP2DS) for magrolimab in combination with rituximab and for magrolimab in combination with rituximab, gemcitabine, and oxaliplatin (R-GemOx).
* To evaluate the efficacy of magrolimab in combination with rituximab in participants with indolent lymphoma and diffuse large B-cell lymphoma (DLBCL) and to evaluate the efficacy of magrolimab in combination with R-GemOx in autologous stem cell transplant (ASCT) ineligible DLBCL participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Phase 1b only: B-cell non-Hodgkin's lymphoma (NHL), relapsed or refractory to standard approved therapies
* DLBCL Phase 2 cohort: De novo or transformed diffuse large B-cell lymphoma (DLBCL) expressing cluster of differentiation (CD) 20, relapsed or refractory to at least 2 prior lines treatment containing anti-CD20 therapy
* Indolent lymphoma Phase 2 cohort: Marginal zone or follicular lymphoma, relapsed or refractory to standard approved therapies
* DLBCL chemotherapy combination cohort: De novo or transformed diffuse large B-cell lymphoma (DLBCL), relapsed or refractory to 1-3 prior lines of treatment
* Adequate performance status and hematological, liver and kidney functions
* Willing to consent to 1 mandatory pre-treatment and 1 on-treatment tumor biopsy

Key Exclusion Criteria:

* Active brain metastases
* Prior allogeneic hematopoietic cell transplantation
* Prior treatment with CD47 or signal regulatory protein alpha (SIRPα) targeting agents
* Second malignancy within the last 3 years
* Known active or chronic hepatitis B or C infection or HIV
* Pregnancy or active breastfeeding
* Prior chimeric antigen receptor (CAR-T) therapy

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (20):
- United States (16):
  - University of Alabama At Birmingham (Uab), Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - National Institutes of Health Clinical Center/ National Cancer Institute, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Washington University School of Medicine Siteman Cancer Center, St Louis, Missouri
  - Levine Cancer Institute, Charlotte, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - St. Vincent's Hospital Melbourne, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- The Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Advani R, Flinn I, Popplewell L, Forero A, Bartlett NL, Ghosh N, Kline J, Roschewski M, LaCasce A, Collins GP, Tran T, Lynn J, Chen JY, Volkmer JP, Agoram B, Huang J, Majeti R, Weissman IL, Takimoto CH, Chao MP, Smith SM. CD47 Blockade by Hu5F9-G4 and Rituximab in Non-Hodgkin's Lymphoma. N Engl J Med. 2018 Nov 1;379(18):1711-1721. doi: 10.1056/NEJMoa1807315. PMID 30380386
- [Background] Advani R, Volkmer JP, Chao MP. CD47 Blockade and Rituximab in Non-Hodgkin's Lymphoma. N Engl J Med. 2019 Jan 31;380(5):497-498. doi: 10.1056/NEJMc1816156. No abstract available. PMID 30699313
- [Background] Mehta A, Popplewell L, Collins GP, Smith S, Flinn I, Bartlett NL, et al. Magrolimab in Combination With Rituximab in Patients With Relapsed or Refractory Indolent Non-Hodgkin Lymphoma: 3-Year Follow-up Results From a Phase 1/2 Trial. Am J Hematol 2022;97:S3-S40.
- [Background] Maakaron J, Asch AS, Popplewell LL, Collins GP, Flinn IW, Ghosh N, et al. Magrolimab in Combination with Rituximab + Chemotherapy in Patients with Relapsed or Refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL). Blood 2022;140 (Supplement 1):3728-3730.
- [Background] Advani R, Bartlett NL, Smith SM, Roschewski M, Popplewell L, Flinn I, et al. Activity of thefirst-in-class anti-CD47 antibody Hu5F9-G4 with rituximab in relapsed/refractory Non-Hodgkin's lymphoma: interim Phase 1b/2 results [Presentation]. 15th International Conference on Malignant Lymphoma (ICML); 2019 18-22 June; Lugano, Switzerland.
- [Background] Advani R, Bartlett NL, Smith SM, Roschewski M, Popplewell L, Flinn I, et al. The first-in-class anti-CD47 antibody Hu5F9-G4 + rituximab induces durable responses in relapsed/refractory DLBCL and indolent lymphoma: Interim Phase 1b/2 results [Abstract]. 15th International Conference on Malignant Lymphoma (ICML); 2019 18-22 June; Lugano, Switzerland.
- [Background] Roschewski M, Advani R, Bartlett NL, Smith SM, Popplewell L, Flinn I, et al. Activity of the first-in-class anti-CD47 antibody Hu5F9-G4 with rituximab in relapsed/refractory Non-Hodgkin's lymphoma: interim Phase 1b/2 results [Presentation]. 24th Congress of the European Hematology Association (EHA); 2019 13-16 June; Amsterdam, Netherlands.
- [Background] Advani R, Bartlett NL, Smith SM, Roschewski M, Popplewell L, Flinn I, et al. The first-in-class anti-CD47 antibody Hu5F9-G4 with rituximab induces durable responses in relapsed/refractory DLBCL and indolent lymphoma: Interim Phase 1b/2 results [Abstract]. 24th Congress of the European Hematology Association (EHA); 2019 13-16 June; Amsterdam, Netherlands.
- [Background] Wang B, Jin D, Cho MM, Takimoto C, Chao M, Agoram B. Magrolimab (Hu5F9-G4, 5F9) Treatment Does Not Alter Rituximab Pharmacokinetics in Patients With Non-Hodgkin's Lymphoma [Poster THU-008]. Eleventh American Conference on Pharmacometrics (ACoP11) Virtual; 2020 09-13 November.
- [Background] Wang B, Jin D, Takimoto C, Chao M, Agoram B. Magrolimab Treatment Does Not Alter Rituximab Pharmacokinetics in Patients with Non-Hodgkin's Lymphoma [Abstract]. Eleventh American Conference on Pharmacometrics (ACoP11) Virtual; 2020 09-13 November.
- [Background] Jin DCY, Wang B, Sikic B, Advani R, Chao M, Takimoto C, et al. Population-Pharmacokinetics of Magrolimab (Hu5F9-G4, 5F9) in Patients With Solid Tumors and Lymphomas [Poster TUE-020]. Eleventh American Conference on Pharmacometrics (ACoP11) Virtual; 2020 09-13 November.
- [Background] Jin DCY, Wang B, Sikic B, Advani R, Chao M, Takimoto C, et al. Population pharmacokinetics of magrolimab (5F9, Hu5F9-G4) in patients with solid tumors and lymphomas [Abstract]. Eleventh American Conference on Pharmacometrics (ACoP11) Virtual; 2020 09-13 November.
- [Derived] Maakaron JE, Asch A, Popplewell L, Collins GP, Flinn IW, Ghosh N, Keane C, Ku M, Mehta A, Roschewski M, Hacohen-Kleiman G, Huo Y, Zhang Y, Renard C, Smith SM, Advani R. Magrolimab plus rituximab with or without chemotherapy in patients with relapsed/refractory diffuse large B-cell lymphoma. Blood Adv. 2024 Nov 26;8(22):5864-5874. doi: 10.1182/bloodadvances.2024013338. PMID 39293083
- [Derived] Mehta A, Popplewell L, Collins GP, Smith SM, Flinn IW, Bartlett NL, Ghosh N, Hacohen-Kleiman G, Huo Y, Su-Feher L, Renard C, Advani R, Roschewski M. Magrolimab plus rituximab in relapsed/refractory indolent non-Hodgkin lymphoma: 3-year follow-up of a phase 1/2 trial. Blood Adv. 2024 Nov 26;8(22):5855-5863. doi: 10.1182/bloodadvances.2024013277. PMID 39213421
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=5F9003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, the United Kingdom, and the United States.
Pre-assignment Details: 209 participants were screened.
Groups:
- Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab: Participants with B-cell non-hodgkin's lymphoma (NHL) received 1 mg/kg magrolimab intravenous (IV) infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 10 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 86.6 months.
- Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 20 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 83.3 months.
- Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11,15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 67.9 months.
- Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 29.2 months.
- Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible diffuse large B-cell lymphoma (DLBCL) participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 30 mg/kg on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. Granulocyte colony stimulating factor (G-CSF) prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
  The maximum duration of treatment was up to approximately 23.2 months.
- Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 45 mg/kg on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
  The maximum duration of treatment was up to approximately 10.8 months.
- Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab: Participants with B-cell indolent NHL (iNHL) (including follicular lymphoma [FL] and marginal zone lymphoma [MZL]) and DLBCL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 59.9 months.
- Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab: Participants with B-cell iNHL (including FL and MZL) and DLBCL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, and 22 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 15.7 months.
- Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab: Participants with B-cell iNHL (including FL and MZL) and DLBCL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11, 15, and 22 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 57.4 months.
- Phase 2 Cohort 4: Magrolimab 30 mg/kg + Rituximab: Participants with DLBCL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each Cycle length was 28 days.
  The maximum duration of treatment was up to approximately 35.3 months.
Period: Overall Study
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab | Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab | Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab | Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab | Phase 2 Cohort 4: Magrolimab 30 mg/kg + Rituximab
Started | 3 | 6 | 13 | 7 | 26 | 7 | 43 | 14 | 31 | 28
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 13 | 7 | 26 | 7 | 43 | 14 | 31 | 28
Not completed — Death | 1 | 3 | 3 | 4 | 12 | 3 | 25 | 10 | 21 | 20
Not completed — Reason Not Specified | 0 | 2 | 8 | 2 | 11 | 4 | 12 | 2 | 7 | 2
Not completed — Consent Withdrawn | 1 | 1 | 2 | 1 | 3 | 0 | 4 | 1 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Study terminated by sponsor | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab intravenous (IV) infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 10 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 86.6 months.
- Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 30 mg/kg on Days 8, 11, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
  The maximum duration of treatment was up to approximately 23.2 months.
- Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab: Participants with B-cell iNHL (including FL and MZL) and DLBCL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 59.9 months.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab | Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab | Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab | Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab | Phase 2 Cohort 4: Magrolimab 30 mg/kg + Rituximab | Total~(N=178)
Number analyzed (Participants) | 3 | 6 | 13 | 7 | 26 | 7 | 43 | 14 | 31 | 28 | 178
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 8 | 4 | 9 | 3 | 21 | 2 | 8 | 8 | 70
  >=65 years | 1 | 1 | 5 | 3 | 17 | 4 | 22 | 12 | 23 | 20 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.8) | 60 (11.3) | 61 (11.4) | 63 (15.2) | 65 (14.4) | 70 (9.5) | 62 (13.2) | 71 (6.7) | 70 (11.5) | 70 (12.4) | 66 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 1 | 10 | 2 | 16 | 4 | 15 | 9 | 67
  Male | 1 | 3 | 8 | 6 | 16 | 5 | 27 | 10 | 16 | 19 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 3 | 2 | 11
  Not Hispanic or Latino | 3 | 5 | 12 | 7 | 24 | 4 | 41 | 14 | 28 | 24 | 162
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 7
  White | 3 | 4 | 10 | 7 | 20 | 5 | 39 | 14 | 28 | 24 | 154
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 3 | 2 | 1 | 0 | 1 | 3 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 13 | 7 | 24 | 7 | 39 | 13 | 28 | 22 | 162
  United Kingdom | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 1 | 3 | 2 | 12
  Australia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Percentage of Participants Experiencing Dose-limiting Toxicities (DLTs) in Antibody Treatment Combination
Description: DLTs refer to toxicities experienced during the first 28 days of study treatment that have been judged to be clinically significant and related to study treatment in participant in Phase 1b. A DLT was defined as any Grade 3 or greater AE that was assessed as related to either magrolimab and/or rituximab that occurred during the 4-week DLT observation period. Any treatment-emergent adverse event (TEAE) that was, in the opinion of the Clinical Trial Steering Committee, of potential clinical significance such that further dosing exposed participants to unacceptable risk, was considered a DLT.
Time Frame: Up to 28 days
Population: The DLT Analysis Set 1 (Antibody Combination) included all enrolled Phase 1b participants in the magrolimab + rituximab cohort who met either of the following criteria:
  * The participant experienced a DLT
  * The participants completed at least 3 infusions of magrolimab and 2 infusions of rituximab.
Measure: Number; unit: percentage of participants
Groups:
- Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 67.9 months.
- Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and beyond in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 29.2 months.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab
Number analyzed (Participants) | 3 | 6 | 13 | 6
percentage of participants | 0 | 16.7 | 15.4 | 16.7

2. Primary Outcome: Phase 1b: Percentage of Participants Experiencing Dose-limiting Toxicities (DLTs) in Chemotherapy Treatment Combination
Description: DLTs refer to toxicities experienced during the first 28 days of study treatment that have been judged to be clinically significant and related to study treatment in participant in Phase 1b. DLT was defined as any Grade 3 or greater AE including Grade 4 hematologic toxicity that does not resolve to Grade 2 and delays initiation of cycle 2 by more than 14 days, Grade 4 febrile neutropenia or associated infections, Grade 4 non-hematologic toxicity that does not resolve or decrease to Grade 2 within 1 week, Grade 4 infusion-related reaction (IRR), and recurrent Grade 3 or greater IRR despite optimal pretreatment regimen that was assessed as related to either magrolimab, rituximab, gemcitabine, or oxaliplatin and occurred during the 4-week DLT observation period. Any TEAE that was, in the opinion of the Clinical Trial Steering Committee, of potential clinical significance such that further dosing exposed participants to unacceptable risk, was considered a DLT.
Time Frame: Up to 28 days
Population: The DLT Analysis Set 2 (Chemotherapy Combination)included all enrolled Phase 1b participants in the magrolimab + rituximab, gemcitabine,and oxaliplatin (R-GemOx) cohort who met either of the following criteria in DLT assessment period:
  * Participants had DLT at any time after initiation of first infusion of magrolimab, rituximab, and gemcitabine or oxaliplatin
  * Participants completed at least 3 infusions of magrolimab, 2 infusions of rituximab, and 1 infusion of gemcitabine and oxaliplatin
Measure: Number; unit: percentage of participants
Groups:
- Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible diffuse large B-cell lymphoma (DLBCL) participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 30 mg/kg on Days 8, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
  The maximum duration of treatment was up to approximately 23.2 months.
- Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 45 mg/kg on Days 8, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
  The maximum duration of treatment was up to approximately 10.8 months.
Arm/Group | Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Number analyzed (Participants) | 5 | 6
percentage of participants | 0 | 16.7

3. Primary Outcome: Percentage of Participants Experiencing Treatment Emergent Adverse Events (TEAEs)
Description: TEAE's were defined as any AEs with an onset date on or after the study drug start date, no later than 30 days after last dose of any study drug or day before initiation of subsequent line of anti-cancer therapy, whichever is earlier, or the AEs leading to the discontinuation of the study drug. An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with use of an investigational product or other protocol imposed intervention, regardless of attribution.
Time Frame: Up to 7.2 years
Population: The Safety Analysis Set included all participants who received at least 1 dose of any study treatment.
Measure: Number; unit: percentage of participants
Groups:
- Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 30 mg/kg on Days 8, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
  The maximum duration of treatment was up to approximately 23.2 months.
- Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab: Participants with B-cell iNHL (including FL and MZL) and DLBCL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 15.7 months.
- Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab: Participants with B-cell iNHL (including FL and MZL) and DLBCL received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Each cycle length was 28 days.
  The maximum duration of treatment was up to approximately 57.4 months.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab | Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab | Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab | Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab | Phase 2 Cohort 4: Magrolimab 30 mg/kg + Rituximab
Number analyzed (Participants) | 3 | 6 | 13 | 7 | 26 | 7 | 43 | 14 | 31 | 28
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 96.2 | 100.0 | 97.7 | 100.0 | 100.0 | 100.0

4. Primary Outcome: Objective Response Rate (ORR) (Complete Response [CR] + Partial Response [PR]) as Defined by the Investigator According to the Lugano Classification for Lymphomas
Description: ORR:CR(complete metabolic response(CMR);complete radiological response(CRR)) or PR(partial metabolic response(PMR);partial radiologic response(PRR)).CMR:PET 5 point-scale(5PS) with 1(no uptake above background,2(uptake≤mediastinum),3(uptake>mediastinum but≤liver)with/without residual mass;no new lesions;no fluorodeoxyglucose (FDG)-avid disease in bone marrow(BM).CRR:target nodes/nodal masses regressed ≤1.5cm in longest transverse diameter of lesion(LDi);no extra lymphatic disease sites;absent non-measured lesions(NMLs);organ enlargement to normal;no new sites;BM morphology normal.PMR:scores 4(uptake moderately>liver),5(uptake markedly>liver,new lesions)with reduced uptake from baseline & residual mass;no new lesion;responding disease at interim/residual disease at end of treatment.PRR:≥50% decrease in sum of perpendicular diameters up to 6 target measurable nodes,extra-nodal sites;absent/normal,regressed,but no increase of NMLs;spleen regressed >50% length beyond normal; no new sites.
Time Frame: Up to 7.3 years
Population: The Efficacy Analysis Set included all enrolled participants who received at least 1 dose of magrolimab. As prespecified in the statistical analysis plan (SAP), the efficacy results were to be reported for Phase 1b and 2 combined per dose and disease type (for both antibody and chemotherapy combinations).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Magrolimab 10 mg/kg + Rituximab (DLBCL): All DLBCL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 10 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
- Magrolimab 10 mg/kg + Rituximab (iNHL): All iNHL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 10 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
- Magrolimab 20 mg/kg + Rituximab (DLBCL): All DLBCL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 20 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
- Magrolimab 20 mg/kg + Rituximab (iNHL): All iNHL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 20 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
- Magrolimab 30 mg/kg + Rituximab (DLBCL): All DLBCL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 30 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
- Magrolimab 30 mg/kg + Rituximab (iNHL): All iNHL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 30 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
- Magrolimab 45 mg/kg + Rituximab (DLBCL): All DLBCL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 45 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
- Magrolimab 45 mg/kg + Rituximab (iNHL): All iNHL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 45 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
- Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 30 mg/kg on Days 8, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 of Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
- Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 45 mg/kg on Days 8, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
Arm/Group | Magrolimab 10 mg/kg + Rituximab (DLBCL) | Magrolimab 10 mg/kg + Rituximab (iNHL) | Magrolimab 20 mg/kg + Rituximab (DLBCL) | Magrolimab 20 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab (DLBCL) | Magrolimab 30 mg/kg + Rituximab (iNHL) | Magrolimab 45 mg/kg + Rituximab (DLBCL) | Magrolimab 45 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Number analyzed (Participants) | 2 | 1 | 6 | 0 | 68 | 30 | 23 | 15 | 26 | 7
percentage of participants | 0 [0.0 to 84.2] | 0 [0.0 to 97.5] | 50.0 [11.8 to 88.2] |  | 20.6 [11.7 to 32.1] | 60.0 [40.6 to 77.3] | 26.1 [10.2 to 48.4] | 33.3 [11.8 to 61.6] | 46.2 [26.6 to 66.6] | 71.4 [29.0 to 96.3]

5. Secondary Outcome: PK Parameter of Magrolimab: AUClast
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration. N = 0 participants for Phase 1b Cohorts 4 and 6, Phase 2 Cohort 3 (DLBCL and iNHL), since PK samples were not collected for Day 1.
Time Frame: Phase 1: Pre-dose (12 hours) and 1 and 24 hours post-dose on Day 1 (Cycle 1 Day 1 [C1D1]); pre-dose and 1, 24, and 72 hours post-dose on Day 8 (C1D8) and Day 29 (C2D1); Phase 2 :Pre-dose (12 hours) on Days 1 (C1D1), 8 (C1D8), and 29 (C2D1)
Population: The Pharmacokinetics (PK) Analysis Set included all participants who received at least 1 dose of study drug and had measurable concentrations of magrolimab from PK blood samples. Participants in the PK Analysis Set with available data were analyzed. The PK data was reported for Phase 2 (antibody combination) as per maintenance dose level and disease type.
Measure: Mean (Standard Deviation); unit: day*micrograms(μg)/milliliters(mL)
Groups:
- Phase 1b Cohort 1: Magrolimab 10 mg/kg (No Loading Dose) + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 10 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 1b Cohort 2: Magrolimab 20 mg/kg (No Loading Dose) + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 20 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 1b Cohort 3: Magrolimab 30 mg/kg (Loading Dose) + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 1b Cohort 4: Magrolimab 45 mg/kg (Loading Dose) + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 1b Cohort 5: Magrolimab 30 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 30 mg/kg on Days 8,15, 22, and 29 of Cycle 1, Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine, and oxaliplatin IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4.
- Phase 1b Cohort 6: Magrolimab 45 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 45 mg/kg on Days 8, 15, 22, and 29 of Cycle 1, Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1.Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine, and oxaliplatin IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4.
- Phase 2 Cohort 1 (DLBCL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab; Phase 2 Cohort 4: Magrolimab 30 mg/ kg (No Loading Dose) + Rituximab: Participants with DLBCL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 2 Cohort 1 (iNHL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab: Participants with B-cell iNHL (including FL and MZL) received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 2 Cohort 2 (DLBCL): Magrolimab 30 mg/ kg (Loading Dose) + Rituximab: Participants with DLBCL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 2 Cohort 2 (iNHL): Magrolimab 30 mg/kg (Loading Dose) + Rituximab: Participants with B-cell iNHL (including FL and MZL) received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 2 Cohort 3 (DLBCL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab: Participants with DLBCL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1.Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 2 Cohort 3 (iNHL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab: Participants with B-cell iNHL (including FL and MZL) and DLBCL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 2 Cohort 3 (iNHL): Magrolimab 20 mg/kg (Loading Dose) + Rituximab: Participants in this group had magrolimab maintenance dose de-escalated from 45 to 20 mg/kg with the identical dosing schedule of maintenance doses by the Clinical Trial Steering Committee (CTSC). Participants with B-cell iNHL (including FL and MZL) received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 20 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 20 mg/kg on Day 11 of Cycle 1.Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg (No Loading Dose) + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg (No Loading Dose) + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg (Loading Dose) + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 1b Cohort 5: Magrolimab 30 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin | Phase 2 Cohort 1 (DLBCL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab | Phase 2 Cohort 1 (iNHL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab | Phase 2 Cohort 2 (DLBCL): Magrolimab 30 mg/ kg (Loading Dose) + Rituximab | Phase 2 Cohort 2 (iNHL): Magrolimab 30 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (DLBCL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (iNHL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (iNHL): Magrolimab 20 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 4: Magrolimab 30 mg/ kg (No Loading Dose) + Rituximab
Number analyzed (Participants) | 3 | 5 | 14 | 8 | 18 | 7 | 18 | 24 | 14 | 2 | 15 | 12 | 1 | 8
day*micrograms(μg)/milliliters(mL)
  Day 1 (Cycle 1, Day 1): number analyzed (Participants) | 1 | 4 | 14 | 0 | 18 | 0 | 11 | 13 | 14 | 2 | 0 | 0 | 1 | 8
  Day 1 (Cycle 1, Day 1) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  |  | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.
  Day 8 (Cycle 1, Day 8): number analyzed (Participants) | 3 | 5 | 14 | 8 | 18 | 7 | 14 | 20 | 14 | 2 | 15 | 12 | 1 | 8
  Day 8 (Cycle 1, Day 8) | 770 (346) | 1810 (426) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | 2300 (280) | 2220 (877) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.
  Day 29 (Cycle 2, Day 1) | 1470 (431) | 4260 (1050) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.

6. Secondary Outcome: PK Parameter of Magrolimab: AUCtau
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval). N = 0 participants for Phase 1b Cohorts 4 and 6, Phase 2 Cohort 3 (DLBCL and iNHL), since PK samples were not collected for Day 1.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed. The PK data was reported for Phase 2 (antibody combination) as per maintenance dose level and disease type.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Groups:
- Phase 1b Cohort 5: Magrolimab 30 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 30 mg/kg on Days 8, 15, 22, and 29 of Cycle 1, Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine, and oxaliplatin IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4.
- Phase 1b Cohort 6: Magrolimab 45 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 45 mg/kg on Days 8, 15, 22, and 29 of Cycle 1, Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine, and oxaliplatin IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4.
- Phase 2 Cohort 1 (iNHL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab: Participants with B-cell iNHL (including FL and marginal zone lymphoma MZL) received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg (No Loading Dose) + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg (No Loading Dose) + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg (Loading Dose) + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 1b Cohort 5: Magrolimab 30 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin | Phase 2 Cohort 1 (DLBCL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab | Phase 2 Cohort 1 (iNHL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab | Phase 2 Cohort 2 (DLBCL): Magrolimab 30 mg/ kg (Loading Dose) + Rituximab | Phase 2 Cohort 2 (iNHL): Magrolimab 30 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (DLBCL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (iNHL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (iNHL): Magrolimab 20 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 4: Magrolimab 30 mg/ kg (No Loading Dose) + Rituximab
Number analyzed (Participants) | 3 | 5 | 14 | 8 | 18 | 7 | 18 | 24 | 14 | 2 | 15 | 12 | 1 | 8
day*μg/mL
  Day 1 (Cycle 1, Day 1): number analyzed (Participants) | 1 | 4 | 14 | 0 | 18 | 0 | 11 | 13 | 14 | 2 | 0 | 0 | 1 | 8
  Day 1 (Cycle 1, Day 1) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  |  | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.
  Day 8 (Cycle 1, Day 8): number analyzed (Participants) | 1 | 5 | 14 | 8 | 18 | 7 | 14 | 20 | 14 | 2 | 15 | 12 | 1 | 8
  Day 8 (Cycle 1, Day 8) | 671 (NA) — Standard deviation cannot be calculated for 1 participant. | 1810 (426) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | 2300 (280) | 2080 (658) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.
  Day 29 (Cycle 2, Day 1): number analyzed (Participants) | 2 | 5 | 14 | 8 | 18 | 7 | 18 | 24 | 14 | 2 | 15 | 12 | 1 | 8
  Day 29 (Cycle 2, Day 1) | 1220 (97.0) | 4260 (1050) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.

7. Secondary Outcome: PK Parameter of Magrolimab: Cmax
Description: Cmax is defined as the maximum observed concentration of drug. N = 0 participants for Phase 1b Cohorts 4 and 6, Phase 2 Cohort 3 (DLBCL and iNHL), since PK samples were not collected for Day 1.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Phase 1b Cohort 4: Magrolimab 45 mg/kg (Loading Dose) + Rituximab: Participants with B-cell NHL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 11, and 22 of Cycle 1 and Days 1, 8, 15, and 22 of Cycle 2 and subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 2 Cohort 2 (DLBCL): Magrolimab 30 mg/ kg (Loading Dose) + Rituximab: Participants with DLBCL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 20 mg/kg on Day 11 of Cycle 1. Participants also received a loading dose of magrolimab 30 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
- Phase 2 Cohort 3 (DLBCL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab: Participants with DLBCL received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 45 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1, 8, 15, and 22 of Cycle 2 and Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg (No Loading Dose) + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg (No Loading Dose) + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg (Loading Dose) + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 1b Cohort 5: Magrolimab 30 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin | Phase 2 Cohort 1 (DLBCL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab | Phase 2 Cohort 1 (iNHL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab | Phase 2 Cohort 2 (DLBCL): Magrolimab 30 mg/ kg (Loading Dose) + Rituximab | Phase 2 Cohort 2 (iNHL): Magrolimab 30 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (DLBCL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (iNHL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (iNHL): Magrolimab 20 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 4: Magrolimab 30 mg/ kg (No Loading Dose) + Rituximab
Number analyzed (Participants) | 3 | 5 | 14 | 8 | 18 | 7 | 18 | 24 | 14 | 2 | 15 | 12 | 1 | 8
μg/mL
  Day 1 (Cycle 1, Day 1): number analyzed (Participants) | 1 | 4 | 14 | 0 | 18 | 0 | 11 | 13 | 14 | 2 | 0 | 0 | 1 | 8
  Day 1 (Cycle 1, Day 1) | 0.619 (NA) — Standard deviation cannot be calculated for 1 participant. | 1.32 (1.31) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  | 0.477 (0.178) | 0.496 (0.353) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. |  |  | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.
  Day 8 (Cycle 1, Day 8): number analyzed (Participants) | 3 | 5 | 14 | 6 | 18 | 7 | 14 | 20 | 14 | 2 | 11 | 9 | 1 | 8
  Day 8 (Cycle 1, Day 8) | 212 (54.6) | 485 (114) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | 924 (170) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | 906 (160) | 567 (75.7) | 542 (188) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | 918 (251) | 904 (414) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.
  Day 29 (Cycle 2, Day 1): number analyzed (Participants) | 3 | 5 | 14 | 5 | 18 | 5 | 18 | 24 | 14 | 2 | 10 | 9 | 1 | 8
  Day 29 (Cycle 2, Day 1) | 330 (123) | 903 (186) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | 1862 (411) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | 2096 (449) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | 1858 (321) | 2186 (615) | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required. | NA (NA) — Data could not be calculated due to multiple concentration values below the level of detection; at least 3 [or 4] quantifiable data points were required.

8. Secondary Outcome: Percentage of Participants Who Developed Anti-Magrolimab Antibodies (ADA)
Time Frame: Up to 4 years
Population: The ADA analysis set included participants with at least one reported ADA result where participants evaluable for ADA incidence were defined as participants with non-missing baseline sample and at least one sample taken after drug administration during the treatment or follow-up observation period that are appropriate for ADA testing (with reportable result). As prespecified in SAP,ADA results were to be reported for Phase 2 (antibody combination) as per maintenance dose level and disease type.
Measure: Number; unit: percentage of participants
Groups:
- Phase 2 Cohort 1 (iNHL): Magrolimab 30 mg/kg (No Loading Dose)+ Rituximab: Participants with B-cell iNHL (including FL and MZL) received 1 mg/kg magrolimab IV infusion of priming dose (over 3 hours) on Day 1 of Cycle 1, followed by weekly maintenance dose of 30 mg/kg magrolimab IV infusion (over 2 hours) on Days 8, 15, and 22 of Cycle 1, followed by Days 1 and 15 of subsequent cycles in combination with rituximab 375 mg/m^2 IV infusion on Days 8, 15, and 22 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Thereafter from Cycle 8 and subsequent cycles, rituximab was administered on Day 1 of every other cycle (on even cycles). Cycle length was 28 days.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg (No Loading Dose) + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg (No Loading Dose) + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg (Loading Dose) + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 1b Cohort 5: Magrolimab 30 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg (Loading Dose) + Rituximab + Gemcitabine + Oxaliplatin | Phase 2 Cohort 1 (DLBCL): Magrolimab 30 mg/kg (No Loading Dose) + Rituximab | Phase 2 Cohort 1 (iNHL): Magrolimab 30 mg/kg (No Loading Dose)+ Rituximab | Phase 2 Cohort 2 (DLBCL): Magrolimab 30 mg/ kg (Loading Dose) + Rituximab | Phase 2 Cohort 2 (iNHL): Magrolimab 30 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (DLBCL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (iNHL): Magrolimab 45 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 3 (iNHL): Magrolimab 20 mg/kg (Loading Dose) + Rituximab | Phase 2 Cohort 4: Magrolimab 30 mg/ kg (No Loading Dose) + Rituximab
Number analyzed (Participants) | 3 | 6 | 14 | 7 | 15 | 6 | 17 | 24 | 13 | 2 | 11 | 3 | 1 | 3
percentage of participants | 0 | 0 | 0 | 0 | 6.7 | 0 | 0 | 0 | 7.7 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR is measured from when first OR is met(CR or PR)until the first date of documented progressive disease[progressive metabolic disease(PMD);progressive radiologic disease(PRD)]while on study prior to start of next line anti-cancer therapy.Participants with no progressive disease were censored at last response assessment date.Response assessment post start of anti-cancer therapy was excluded from derivation.OR defined in outcome measure 4.PMD:scores 4(uptake moderately>liver),5(uptake markedly>liver,new lesions)with increased uptake from baseline;new FDG-avid foci consistent with lymphoma rather than another etiology;new or recurrent FDG-avid foci in BM.PRD:LDi >1.5 cm;≥ 50% increase from cross product of LDi & perpendicular diameter(PPD);increase in LDi or shortest axis perpendicular to LDi(SDi) of 0.5 cm for lesions ≤ 2 & 1 cm for lesions >2 cm;spleen increased by >50% in length beyond normal;new or recurrent splenomegaly,BM involved;new lesions;progression of pre-existing lesions.
Time Frame: Up to 7.3 years
Population: Participants in the Efficacy Analysis Set with an objective response (CR + PR) and those who had objective response without a subsequent event of disease progression/death were analyzed. As prespecified in the SAP, the efficacy results were to be reported for Phase 1b and 2 combined per dose and disease type (for both antibody and chemotherapy combinations).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Magrolimab 10 mg/kg + Rituximab (iNHL):: All iNHL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 10 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
Arm/Group | Magrolimab 10 mg/kg + Rituximab (DLBCL) | Magrolimab 10 mg/kg + Rituximab (iNHL): | Magrolimab 20 mg/kg + Rituximab (DLBCL) | Magrolimab 20 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab (DLBCL) | Magrolimab 30 mg/kg + Rituximab (iNHL) | Magrolimab 45 mg/kg + Rituximab (DLBCL) | Magrolimab 45 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Number analyzed (Participants) | 0 | 1 | 3 | 0 | 14 | 18 | 6 | 5 | 12 | 5
months |  | NA [NA to NA] — The median, lower, and upper limit of 95% confidence interval (CI) were not estimable due to insufficient number of events. | NA [3.9 to NA] — The median and upper limit of 95% CI were not estimable due to insufficient number of events. |  | 5.5 [3.5 to 22.3] | 15.9 [5.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | 21.2 [1.8 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | 11.3 [3.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | NA [2.0 to NA] — The median and upper limit of 95% CI were not estimable due to insufficient number of events. | 18.0 [4.7 to NA] — The upper limit of 95% CI were not estimable due to insufficient number of events.

10. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is measured from dose initiation until the first date of objectively documented disease progression (PMD; PRD) or death while on study prior to start of the subsequent line of anti-cancer therapy. Participants who do not have progressive disease & not died were censored at last response assessment date.Response assessments after initiation of the subsequent line of anti-cancer therapy will be excluded from derivation. PMD: scores 4 (uptake moderately > liver), 5 (uptake markedly > liver, new lesions) with increased uptake from baseline; new FDG-avid foci consistent with lymphoma rather than another etiology; new or recurrent FDG-avid foci in BM. PRD: LDi >1.5 cm; ≥ 50% increase from cross product of LDi & PPD; increase in LDi or SDi of 0.5 cm for lesions ≤ 2 & 1 cm for lesions >2 cm; spleen increased by >50% in length beyond normal; new or recurrent splenomegaly, BM involvement; new lesions; progression of pre-existing lesions. KM estimates of median was reported.
Time Frame: Up to 7.3 years
Population: Participants in the efficacy analysis set with available data were analyzed. As prespecified in the SAP, the efficacy results were to be reported for Phase 1b and 2 combined per dose and disease type (for both antibody and chemotherapy combinations).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin: Autologous stem cell transplant (or transplantation) ineligible DLBCL participants received 1 mg/kg magrolimab IV infusion priming dose (over 3 hours) on Day 1 of Cycle 1, followed by maintenance dose of 45 mg/kg on Days 8, 15, 22, and 29 of Cycle 1; Days 1, 8, 15, and 22 of Cycle 2 followed by Days 1 and 15 of subsequent cycles. The cycle length was 28 days. Rituximab 375 mg/m^2 IV infusion was administered on Days 8, 15, 22, and 29 of Cycle 1, followed by 1 dose on Day 1 for Cycles 2 to 6. Participants also received a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1.Thereafter from Cycle 8 and beyond, rituximab was administered on Day 1 of every other cycle (on even cycles). Gemcitabine 1000 mg/m^2 and oxaliplatin 100 mg/m^2 IV infusion were administered as on Days 11 and 23 of Cycle 1 and Days 2 and 15 of Cycles 2 to 4. G-CSF prophylaxis was administered with gemcitabine and oxaliplatin treatment (Cycles 1-4). Allopurinol 300 mg orally daily was administered for the first cycle only.
Arm/Group | Magrolimab 10 mg/kg + Rituximab (DLBCL) | Magrolimab 10 mg/kg + Rituximab (iNHL) | Magrolimab 20 mg/kg + Rituximab (DLBCL) | Magrolimab 20 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab (DLBCL) | Magrolimab 30 mg/kg + Rituximab (iNHL) | Magrolimab 45 mg/kg + Rituximab (DLBCL) | Magrolimab 45 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Number analyzed (Participants) | 2 | 1 | 6 | 0 | 68 | 30 | 23 | 15 | 26 | 7
months | 1.6 [1.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — The median, lower, and upper limit of 95% CI was not estimable due to insufficient number of events. | 5.6 [1.2 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. |  | 1.8 [1.6 to 2.1] | 7.5 [5.5 to 23.9] | 2.1 [1.6 to 3.6] | 5.5 [1.8 to 13.0] | 3.9 [2.3 to 11.1] | 20.3 [0.5 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events.

11. Secondary Outcome: Overall Survival (OS)
Description: OS is measured from dose initiation until death.
Time Frame: Up to 7.3 years
Population: Participants in the Efficacy Analysis Set with available were analyzed. As prespecified in the SAP, the efficacy results were to be reported for Phase 1b and 2 combined per dose and disease type (for both antibody and chemotherapy combinations).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Magrolimab 10 mg/kg + Rituximab (iNHL): All IL participants in Phases 1b and 2, antibody combination arms who received a maintenance dose of 10 mg/kg magrolimab IV infusion in combination with rituximab 375 mg/m^2 IV infusion.
Arm/Group | Magrolimab 10 mg/kg + Rituximab (DLBCL) | Magrolimab 10 mg/kg + Rituximab (iNHL) | Magrolimab 20 mg/kg + Rituximab (DLBCL) | Magrolimab 30 mg/kg + Rituximab (DLBCL) | Magrolimab 20 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab (iNHL) | Magrolimab 45 mg/kg + Rituximab (DLBCL) | Magrolimab 45 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Number analyzed (Participants) | 2 | 1 | 6 | 0 | 68 | 30 | 23 | 15 | 26 | 7
months | 13.9 [NA to NA] — The lower and upper limit of 95% CI were not estimable due to insufficient number of events. | NA [NA to NA] — The median, lower and upper limit of 9,5% CI were not estimable due to insufficient number of events. | 32.2 [2.3 to NA] — The upper-limit of 95% CI were not estimable due to insufficient number of events. |  | 8.5 [5.8 to 11.3] | NA [62.9 to NA] — The median and upper-limit of 95% CI were not estimable due to insufficient number of events. | 14.0 [3.4 to 17.4] | 23.7 [3.8 to NA] — The upper-limit of 95% CI were not estimable due to insufficient number of events. | 41.4 [6.1 to NA] — The upper-limit of 95% CI were not estimable due to insufficient number of events. | NA [0.5 to NA] — The median and upper-limit of 95% CI were not estimable due to insufficient number of events.

12. Secondary Outcome: Time to Progression (TTP)
Description: TTP is measured from dose initiation until the first date of objectively documented progressive disease criteria while on study prior to start of next line anti-cancer therapy. Participants with no progressive disease were censored at last response assessment date. Response assessment post start of anti-cancer therapy was excluded from derivation. PMD: scores 4 (uptake moderately > liver), 5 (uptake markedly > liver, new lesions) with increased uptake compared with baseline; new FDG-avid foci consistent with lymphoma rather than another etiology; new or recurrent FDG-avid foci in bone marrow. PRD: LDi >1.5 cm; = 50% increase from cross product of LDi and PPD; increase in LDi or SDi of 0.5 cm for lesions =1.5 cm and 1 cm for lesions >2 cm; spleen increased by >50% in length beyond normal; new or recurrent splenomegaly, bone marrow involvement; new lesions; progression of pre-existing lesions. Kaplan-meier (KM) estimates of median was reported.
Time Frame: Up to 7.3 years
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab 10 mg/kg + Rituximab (DLBCL) | Magrolimab 10 mg/kg + Rituximab (iNHL) | Magrolimab 20 mg/kg + Rituximab (DLBCL) | Magrolimab 20 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab (DLBCL) | Magrolimab 30 mg/kg + Rituximab (iNHL) | Magrolimab 45 mg/kg + Rituximab (DLBCL) | Magrolimab 45 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Number analyzed (Participants) | 2 | 1 | 6 | 0 | 68 | 30 | 23 | 15 | 26 | 7
months | 1.6 [1.4 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — The median, lower, and upper limit of 95% CI was not estimable due to insufficient number of events. | 5.6 [1.2 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. |  | 1.8 [1.7 to 2.1] | 7.9 [5.5 to 23.9] | 2.0 [1.6 to 4.3] | 5.6 [1.8 to 13.0] | 3.9 [2.3 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events. | 20.3 [6.6 to NA] — The upper limit of 95% CI was not estimable due to insufficient number of events.

13. Secondary Outcome: ORR (CR + PR) Defined by the Investigator According to the Lymphoma Response to Immunomodulatory Therapy Criteria for Lymphomas
Description: Objective response is defined as complete response or partial response determined by LYRIC criteria. ORR:CR[CMR;CRR] or PR[PMR;PRR].CMR:PET 5 PS with 1(no uptake above background,2(uptake≤mediastinum),3(uptake>mediastinum but≤liver)with/without residual mass;no new lesions;no FDG-avid disease in BM.CRR:target nodes/nodal masses regressed to ≤1.5cm in LDi;no extralymphatic disease sites;absent NMLs;organ enlargement to normal;no new sites;BM morphology normal.PMR:scores 4(uptake moderately>liver),5(uptake markedly>liver,new lesions)with reduced uptake from baseline and residual mass;no new lesion;responding disease at interim/residual disease at end of treatment.PRR: ≥50% decrease in sum of product of perpendicular diameters up to 6 target measurable nodes,extra-nodal sites;absent/normal,regressed,but no increase of NMLs;spleen regressed >50% in length beyond normal;no new sites.
Time Frame: Up to 7.3 years
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab 10 mg/kg + Rituximab (DLBCL) | Magrolimab 10 mg/kg + Rituximab (iNHL) | Magrolimab 20 mg/kg + Rituximab (DLBCL) | Magrolimab 20 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab (DLBCL) | Magrolimab 30 mg/kg + Rituximab (iNHL) | Magrolimab 45 mg/kg + Rituximab (DLBCL) | Magrolimab 45 mg/kg + Rituximab (iNHL) | Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin
Number analyzed (Participants) | 2 | 1 | 6 | 0 | 68 | 30 | 23 | 15 | 26 | 7
percentage of participants | 0 [0.0 to 84.2] | 0 [0.0 to 97.5] | 50.0 [11.8 to 88.2] |  | 22.1 [12.9 to 33.8] | 60.0 [40.6 to 77.3] | 26.1 [10.2 to 48.4] | 33.3 [11.8 to 61.6] | 46.2 [26.6 to 66.6] | 71.4 [29.0 to 96.3]

ADVERSE EVENTS:
Time Frame: Adverse event: Up to 7.2 years; All-cause mortality: Up to 7.3 years
Description: Adverse Events: The Safety Analysis Set included all enrolled patients who receive at least 1 dose of any study drug.
  All-cause mortality: The Enrolled Analysis Set included all enrolled patients.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab | Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab | Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab | Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab | Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin | Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab | Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab | Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab | Phase 2 Cohort 4: Magrolimab 30 mg/kg + Rituximab
All-Cause Mortality (participants affected / at risk) | 1/3 | 4/6 | 5/13 | 4/7 | 12/26 | 3/7 | 26/43 | 10/14 | 22/31 | 21/28
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6 | 6/13 | 1/7 | 21/26 | 5/7 | 19/43 | 9/14 | 21/31 | 11/28
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 13/13 | 7/7 | 25/26 | 7/7 | 42/43 | 14/14 | 31/31 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab (N=3) | Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab (N=6) | Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab (N=13) | Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab (N=7) | Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin (N=26) | Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin (N=7) | Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab (N=43) | Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab (N=14) | Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab (N=31) | Phase 2 Cohort 4: Magrolimab 30 mg/kg + Rituximab (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retroperitoneal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Death, not otherwise specified (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 4 | 1 | 3 | 2 | 5 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Rituximab (N=3) | Phase 1b Cohort 2: Magrolimab 20 mg/kg + Rituximab (N=6) | Phase 1b Cohort 3: Magrolimab 30 mg/kg + Rituximab (N=13) | Phase 1b Cohort 4: Magrolimab 45 mg/kg + Rituximab (N=7) | Phase 1b Cohort 5: Magrolimab 30 mg/kg + Rituximab + Gemcitabine + Oxaliplatin (N=26) | Phase 1b Cohort 6: Magrolimab 45 mg/kg + Rituximab + Gemcitabine + Oxaliplatin (N=7) | Phase 2 Cohort 1: Magrolimab 30 mg/kg + Rituximab (N=43) | Phase 2 Cohort 2: Magrolimab 30 mg/kg + Rituximab (N=14) | Phase 2 Cohort 3: Magrolimab 45 mg/kg + Rituximab (N=31) | Phase 2 Cohort 4: Magrolimab 30 mg/kg + Rituximab (N=28)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 0 | 20 | 3 | 15 | 4 | 10 | 11
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 2
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 1 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0 | 4 | 2 | 8 | 1 | 6 | 5
Red blood cell agglutination (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 1 | 13 | 2 | 5 | 2 | 5 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 3 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Iritis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 6 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3 | 1 | 7 | 2 | 2 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 10 | 0 | 8 | 1 | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 8 | 2 | 15 | 5 | 12 | 0 | 6 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 7 | 1 | 13 | 5 | 15 | 4 | 10 | 6
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 5 | 1 | 7 | 3 | 12 | 1 | 8 | 4
Asthenia (General disorders) | 1 | 1 | 0 | 1 | 5 | 1 | 2 | 0 | 5 | 0
Catheter site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Catheter site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site vesicles (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Chills (General disorders) | 2 | 4 | 5 | 2 | 6 | 2 | 15 | 6 | 7 | 5
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 5 | 9 | 4 | 18 | 5 | 18 | 5 | 11 | 9
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Infusion site swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2 | 1 | 5 | 1 | 5 | 2 | 3 | 5
Pain (General disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 3
Peripheral swelling (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 5 | 3 | 7 | 2 | 14 | 2 | 11 | 8
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 4 | 0 | 3 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Infected bite (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 3 | 4 | 1 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 5 | 0 | 3 | 2 | 9 | 0 | 6 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 0 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0 | 3 | 1 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 3 | 1 | 7 | 0 | 4 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 | 7 | 4 | 12 | 2 | 20 | 2 | 11 | 11
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 4 | 1 | 1 | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 4 | 1 | 1 | 1 | 2 | 1
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 5
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cd4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haptoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Immunoglobulins decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 4 | 2 | 1 | 0 | 3 | 0 | 1 | 4
Platelet count decreased (Investigations) | 0 | 1 | 2 | 1 | 9 | 2 | 6 | 2 | 2 | 6
Total lung capacity decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 2 | 1 | 2 | 2 | 1 | 0 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 6 | 2 | 6 | 4 | 10 | 2 | 7 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 4 | 1 | 2 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 8 | 0 | 3 | 0 | 4 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 5 | 1 | 2 | 1 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 1 | 3 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 6 | 0 | 2 | 0 | 2 | 3
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 0 | 0 | 2 | 5 | 4 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 7 | 2 | 2 | 4 | 10 | 3 | 6 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 2 | 0 | 4 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 1 | 1 | 6 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 3 | 0 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 5 | 1 | 3 | 2 | 4 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral microangiopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 2 | 1 | 6 | 5 | 3 | 3 | 5 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 5 | 9 | 4 | 8 | 3 | 25 | 1 | 7 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypogeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Vibratory sense increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 3 | 0 | 1 | 1 | 4 | 0 | 2 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 6 | 1 | 5 | 4 | 17 | 0 | 8 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 3 | 2 | 8 | 4 | 13 | 3 | 10 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 3 | 4 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1 | 2 | 0 | 3 | 1 | 6 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 3 | 0 | 2 | 1 | 1 | 2
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1 | 2 | 3 | 0 | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3 | 2 | 0 | 8 | 0 | 2 | 2
Purpura senile (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1 | 0 | 6 | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 4 | 2 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 1 | 3 | 1 | 6 | 3 | 6 | 2 | 4 | 5
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Varicose vein (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT02953509/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT02953509/SAP_001.pdf